CLINICAL TRIAL: NCT03852173
Title: Process and Outcome Evaluation of an Intervention to Increase the Water Consumption of Elementary School Children in Lower Austria - a Pilot Study
Brief Title: Effects of a School-based Intervention to Increase the Water Consumption in Elementary School Children
Acronym: H2NOE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danube University Krems (Other)
Collaborators: Lower Austrian Health and Social Fund (Unknown); Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ursula Griebler, Principal investigator, Danube University Krems
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H2NOE-Wasserschule
Record Dates: First submitted 2019-02-19; First posted 2019-02-25 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Water Consumption; Drinking Behavior
Keywords: Child; Health promotion; longitudinal studies; Surveys and Questionnaires; beverages; Water/administration & dosage; Austria; Program evaluation; Students/statistics & numerical data; Food Preferences; Follow-Up Studies; school setting; behavioural change
MeSH Terms: conditions — Drinking Behavior; Food Preferences

STUDY DESIGN:
Intervention Model Description: Intervention versus no intervention
Who Masked: Participant
Masking Description: Participants in the control group are not aware that they serve as control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group "Wasserschulen" (Experimental): Schools receive refillable drinking bottles for all school children and drying racks for each classroom. Schools receive special project educational material and informational material and one training session for teachers. The intervention will be implemented during one school year (2018/2019), but schools can use the material and bottles also after ending of the intervention period.
  Interventions: Behavioral: Wasserschulen
- Control group (No Intervention): No intervention (usual education). Schools do not receive any project material. Schools got the information that they are part of a study on drinking and eating habits of third grade elementary school children.

INTERVENTIONS:
Behavioral: Wasserschulen — Schools receive following materials and trainings:
  * one training sessions for teachers (at the beginning of the intervention)
  * refillable water bottles for each school student
  * drying rack for water bottles for each classroom
  * educational material for each class and for school events
  * informational material for parents
  Arms: Intervention group "Wasserschulen"

SUMMARY:
The purpose of this controlled intervention study is to evaluate the effectiveness of a school-based intervention aiming at increasing the water consumption in elementary school children. The intervention schools received refillable water bottles and drying racks for all school children as well as educational material. The focus of the intervention is the promotion of drinking tap water.

DETAILED DESCRIPTION:
This pilot project, called "H2NOE-Wasserschulen" (Water Schools in Lower Austria), aims to increase the water consumption of school children in elementary schools, to raise awareness of water drinking in children, parents and school teachers and to promote water drinking in Lower Austria in general.

By increasing the consumption of water, the consumption of sugar-sweetened beverages may decrease and in the long run may have a positive impact on children's body weight and tooth status.

All intervention schools receive refillable water bottles for each school child and drying racks for each classroom. Furthermore, in each school an information session for all school teachers is held and the teachers receive prepared educational material. The control schools do not receive the water bottles nor the educational material.

For the study, the investigators recruited 22 intervention schools and 32 control schools. Outcomes will be measured by paper and pencil questionnaires of school children at third grade of participating elementary schools in Lower Austria and with online questionnaires of teachers at baseline, at the end of the intervention (after one school year/June 2019) and at the one-year follow-up (after two school years/June 2020).

For process evaluation outcomes, the investigators will carry out focus group discussions with a subsample of school children and teachers and include questions in the respective questionnaires for school children, teachers and school headmasters. Parents will have the possibility to give feedback online.

ELIGIBILITY:
For the intervention schools:

Inclusion criteria:

* elementary school in Niederösterreich (Upper Austria, a province of Austria)
* no juice provided with the school milk programme

For the school children taking part in the survey:

Inclusion criteria:

* school children in third class of elementary school (at baseline)
* written declaration of consent by a parent/guardian

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1485 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Change in water consumption of school children (from baseline to post-intervention and follow-up) | baseline, end of intervention (after one school year, 9 months), follow-up (after two school years, 21 months)
  consumption of tap water, in number of glasses (with 1 glass defined as 200 mL) per day/ during school time (self-report)
Change of attitude of school children towards drinking water (from baseline to post-intervention and follow-up) | baseline, end of intervention (after one school year, 9 months), follow-up (after two school years, 21 months)
  preference for water and sugar-sweetened beverages (measured as agreement to various statements regarding water and sugar-sweetened beverage consumption with 5 likert-scale answer categories: yes, that's right; yes, mostly; no, mostly not; no, not true; I don't know)

SECONDARY OUTCOMES:
Change in beverage consumption of school children (from baseline to post-intervention and follow-up) | baseline, end of intervention (after one school year, 9 months), follow-up (after two school years, 21 months)
  consumption of tap water, mineral water, fruit- and herbal tea, milk and cacao, soft drinks (lemonade, cola and iced tea), juice and juice with water; in number of glasses (with 1 glass defined as 200 mL) for the last 24h
Change in food consumption of school children (from baseline to post-intervention and follow-up) | baseline, end of intervention (after one school year, 9 months), follow-up (after two school years, 21 months)
  consumption of fruit and berries; vegetables (raw or cooked); sweets, chocolate or ice-cream; soft drinks (lemonade, cola and iced tea); fast food (french fries, chicken nuggets, pizza, McDonald's, sausages); salty snacks (crisps, popcorn, salted pretzel sticks); frequency of consumption during a normal week, when thinking of the last weeks
Change in breakfast consumption of school children (from baseline to post-intervention and follow-up) | baseline, end of intervention (after one school year, 9 months), follow-up (after two school years, 21 months)
  frequency of eating breakfast during school days and on the weekend
Parameters of process evaluation (implementation dose) | end of intervention (after one school year, 9 months)
  frequency of addressing the topic water during regular lessons, implementation of classroom rules for water drinking, extent of water bottle use of school children; by online questionnaire (all teachers from intervention schools); extent of water bottle use, by paper and pencil questionnaire (all school children from intervention schools); number of interventional material distributed in school; by online questionnaire (all headmasters from intervention schools)
Parameters of process evaluation (implementation fidelity) | end of intervention (after one school year, 9 months)
  implementation of classroom rules for water drinking; extent of information for parents; by online questionnaire (all teachers from intervention schools)
Parameters of process evaluation (implementation reach) | end of intervention (after one school year, 9 months)
  proportion of classes that implemented the intervention, information about intervention on the school homepage, number of interventional material distributed in school; by online questionnaire (all headmasters from intervention schools); extent of information for parents; by online questionnaire (all teachers from intervention schools)
Parameters of process evaluation (acceptance) | end of intervention (after one school year, 9 months)
  focus group discussions with a subset of school children, teachers and school headmasters

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Griebler, PhD, MPH, Principal Investigator — Danube University Krems
Locations (1):
- Lower Austrian Health and Social Fund, Sankt Pölten, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Griebler U, Titscher V, Weber M, Affengruber L. Evaluation of the 'H2NOE Water Schools' programme to promote water consumption in elementary schoolchildren: a non-randomised controlled cluster trial. Public Health Nutr. 2022 Jan;25(1):159-169. doi: 10.1017/S1368980021003438. Epub 2021 Aug 13. PMID 34384513